CLINICAL TRIAL: NCT05865704
Title: Childbirth-related Post-traumatic Stress Disorder in Switzerland and Understanding Its Relations With Depression, Health Care Renunciation, Coparenting and Parental Burnout: The Swiss Cohort on Traumatic Childbirth and Health
Brief Title: Childbirth-related Post-traumatic Stress Disorder in Switzerland: The Swiss Cohort on Traumatic Childbirth and Health
Acronym: SwiTCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antje Horsch, Prof., Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2022-284
Record Dates: First submitted 2023-03-21; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: childbirth; posttraumatic stress disorder; birth trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Birth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the prevalence of Childbirth post-traumatic stress disorder (CB-PTSD) and Childbirth post-traumatic stress symptom (CB-PTSS) in Switzerland, and to analyze the psychological, medical, and social factors linked with CB-PTSD and CB-PTSS, whether they are antecedent factors or further consequences.

The main questions it aims to answer are :

* The prevalence of CB-PTSS and CB-PTSD in Switzerland, for both mothers and partners (Primary outcome)
* The risk and protective factors of CB-PTSD and CB-PTSS (Secondary outcome)
* The impact of CB-PTSD and CB-PTSS on the marital and co-parental adjustment and the bonding with the infant (Secondary outcome)
* The role of the childbirth experience on the triggering of CB-PTSD and CB-PTSS, including emotional and affective aspects (Secondary outcome)
* The social and economic determinants of CB-PTSD and CB-PTSS, including, for example, social support and religion (Secondary outcome)

Participants will fill up surveys at four time points:

* T1, during the third trimester of pregnancy
* T2, at 6 to 12 weeks post-partum
* T3, at 6 months post-partum
* T4, at 12 months post-partum

DETAILED DESCRIPTION:
Study design:

The present study consists of a longitudinal cohort study with surveys at four time points:

* T1: Third trimester of pregnancy: including risk and protective factors for PTSD such as antenatal stress, mother-partner relationships, social support, current anxiety and depression, and history of mental health issues and treatments. Sociodemographic information is also collected at this time.
* T2: 6-12 weeks postpartum: focusing on delivery conditions and its consequences with an extra focus on determining whether childbirth included eligible traumatic events such as e.g. emergency C-section, forceps, vacuum. The survey also investigates immediate PTSD onsets and other short-term outcomes such as early co-parenting quality and parent-infant bonding.
* T3: 6 months postpartum: including reassessment of CB-PTSD since CB-PTSD occurring more than 6 months after the traumatic event represents the "delayed PTSD" subtype.
* T4: 12 months postpartum: in order to identify the prevalence of delayed CB-PTSD, or of persistent/recurrent perinatal depression, to assess parent healthcare renunciation, as well as couple relationship quality/satisfaction and co-parenting quality.

Participants enter the SwiTCH study preferably at T1, but inclusion at T2 is also possible in order to maximize recruitment. The participants included at t2 will fill the sociodemographic and history of mental health surveys at T2 instead of T1.

Study population:

The inclusion criteria for mothers is being pregnant in the third pregnancy trimester and being above 16 years, or being between 6 to 12 weeks postpartum and above 16 years. Partners are recruited based on the inclusion criteria for mothers. Additionally, they must be 16 years old or older.

All participants are asked to sign a written consent (and if applicable, legal representatives for adolescents aged over 16 years old).

ELIGIBILITY:
Inclusion Criteria:

* Women being pregnant in the third pregnancy trimester, or being between 6 to 12 weeks postpartum. Partners are recruited base on the inclusion criteria for mothers.

Exclusion Criteria:

* N/A.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population speaks French since the surveys are in French. The population is recruited in the French speaking part of Switzerland (Vaud, Neuchâtel, Geneva, Friburg, Wallis) in Lausanne University Hospital, in regional hospitals, and at independant healthcare professionals (such as midwifes, gynecologist, doulas...)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of childbirth trauma in mother and partner | 6-12 weeks postpartum
  Measure of the extent to which the birth is perceived as traumatic
Prevalence of childbirth Posttraumatic Stress Disorder (PTSD) and childbirth Postraumatic Stress Symptoms (PTSS) | 6-12 weeks postpartum
  Childbirth-related PTSD and PTSS is assessed with the City Birth Trauma Scale (City BiTS).
Prevalence of childbirth Posttraumatic Stress Disorder (PTSD) and childbirth Postraumatic Stress Symptoms (PTSS) | 6 months postpartum
  Childbirth-related PTSD and PTSS is assessed with the City Birth Trauma Scale (City BiTS).
Prevalence of childbirth Posttraumatic Stress Disorder (PTSD) and childbirth Postraumatic Stress Symptoms (PTSS) | 12 months postpartum
  Childbirth-related PTSD and PTSS is assessed with the City Birth Trauma Scale (City BiTS).

SECONDARY OUTCOMES:
Risk factors of CB-PTSD : History of mental health issues (Mother) | Baseline (Third trimester of pregnancy)
  History of mental health issues/treatment, 4 items
Risk factors of CB-PTSD : History of mental health issues (Partner) | Baseline (Third trimester of pregnancy)
  History of mental health issues/treatment, 4 items
Risk factors of CB-PTSD : Anxiety (Mother) | Baseline (Third trimester of pregnancy)
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Risk factors of CB-PTSD : Anxiety (Partner) | Baseline (Third trimester of pregnancy)
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Risk factors of CB-PTSD : Depression (Mother) | Baseline (Third trimester of pregnancy)
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Risk factors of CB-PTSD : Depression (Patner) | Baseline (Third trimester of pregnancy)
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Risk factors of CB-PTSD : Fear of childbirth I (Mother) | Baseline (Third trimester of pregnancy)
  Fear of childbirth, 1 item
Risk factors of CB-PTSD : Fear of childbirth (Partner) | Baseline (Third trimester of pregnancy)
  Fear of childbirth, 1 item
Risk factors of CB-PTSD : Fear of childbirth II (Mother) | Baseline (Third trimester of pregnancy)
  Fear of Childbirth Questionnaire (FCQ; Slade et al., 2022), 20 items scored on a 4-point scale
Risk factors of CB-PTSD : Antenatal Stress (Mother) | Baseline (Third trimester of pregnancy)
  Antenatal Perceived Stress Inventory (APSI (Razurel et al., 2014), 12 items scored on a 5-point scale
Risk factors of CB-PTSD : Previous trauma (Mother) | Baseline (Third trimester of pregnancy)
  Previous birth trauma, 1 item
Risk factors of CB-PTSD : Previous trauma (Partner) | Baseline (Third trimester of pregnancy)
  Previous birth trauma, 1 item
Risk factors of CB-PTSD : Previous birth trauma (Mother) | Baseline (Third trimester of pregnancy)
  Previous birth trauma, 1 item
Risk factors of CB-PTSD : Previous birth trauma (Partner) | Baseline (Third trimester of pregnancy)
  Previous birth trauma, 1 item
Risk factors of CB-PTSD : Prenatal attachment (Mother) | Baseline (Third trimester of pregnancy)
  Prenatal Attachment Inventory (PAI; Jurgens et al., 2010), 21 items scored on a 4-point scale
Risk factors of CB-PTSD : Relationship satisfaction (Mother) | Baseline (Third trimester of pregnancy)
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Risk factors of CB-PTSD : Relationship satisfaction (Partner) | Baseline (Third trimester of pregnancy)
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Risk factors of CB-PTSD : Social Support (Mother) | Baseline (Third trimester of pregnancy)
  Modified Medical Outcomes Study Social Support Survey (mMOS-SS; Moser et al., 2012), 8 items scored on a 5-point scale
Risk factors of CB-PTSD : Social Support (Partner) | Baseline (Third trimester of pregnancy)
  Modified Medical Outcomes Study Social Support Survey (mMOS-SS; Moser et al., 2012), 8 items scored on a 5-point scale
Consequences of CB-PTSD : Anxiety (Mother) | 6-12 weeks postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Anxiety (Partner) | 6-12 weeks postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Mother) | 6-12 weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Partner) | 6-12 weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Mother-infant bonding I (Mother) | 6-12 weeks postpartum
  Postpartum Bonding Questionnaire (PPBQ; Demanche et al., 2021), 25 items scored on a 5-point scale
Consequences of CB-PTSD : Mother-infant bonding II (Mother) | 6-12 weeks postpartum
  Parent-Infant Bonding Scale (MIBS; Bienfait et al., 2017), 8 items scored on a 4-point scale
Consequences of CB-PTSD : Father-infant bonding (Partner) | 6-12 weeks postpartum
  Parent-Infant Bonding Scale (MIBS; Bienfait et al., 2017), 8 items scored on a 4-point scale
Consequences of CB-PTSD : Relationship satisfaction (Mother) | 6-12 weeks postpartum
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Consequences of CB-PTSD : Relationship satisfaction (Partner) | 6-12 weeks postpartum
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Consequences of CB-PTSD : Coparenting (Mother) | 6-12 weeks postpartum
  Coparenting Relationship Scale (CRS; Favez et al., 2021), 35 items scored on a 7-point scale
Consequences of CB-PTSD : Coparenting (Partner) | 6-12 weeks postpartum
  Coparenting Relationship Scale (CRS; Favez et al., 2021), 35 items scored on a 7-point scale
Consequences of CB-PTSD : Parenting self-efficacy (Mother) | 6-12 weeks postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP-SE; Schneider et al., 2019), 20 items scored on a 4-point scale
Consequences of CB-PTSD : Parenting self-efficacy (Partner) | 6-12 weeks postpartum
  Perceived Maternal Parenting Self-Efficacy (PMP-SE; Schneider et al., 2019), 20 items scored on a 4-point scale
Consequences of CB-PTSD : Healthcare renunciation (Mother) | 6-12 weeks postpartum
  Healthcare renunciation, 3 items
Consequences of CB-PTSD : Healthcare renunciation (Partner) | 6-12 weeks postpartum
  Healthcare renunciation, 3 items
Consequences of CB-PTSD : Anxiety (Mother) | 6 months postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Anxiety (Partner) | 6 months postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Mother) | 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Partner) | 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Mother-infant bonding (Mother) | 6 months postpartum
  Postpartum Bonding Questionnaire (PPBQ; Demanche et al., 2021), 25 items scored on a 5-point scale
Consequences of CB-PTSD : Support from neighborhood (Mother) | 6 months postpartum
  Perceived Neighborhood Social Cohesion (P-NSC; Dupuis et al., 2017), 9 items scored on a 7-point scale
Consequences of CB-PTSD : Support from neighborhood (Partner) | 6 months postpartum
  Perceived Neighborhood Social Cohesion (P-NSC; Dupuis et al., 2017), 9 items scored on a 7-point scale
Consequences of CB-PTSD : Anxiety (Mother) | 12 months postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Anxiety (Partner) | 12 months postpartum
  Hospital Anxiety and Depression Scale (HADS; Untas et al., 2009), 7 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Mother) | 12 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Depression (Partner) | 12 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS; Guedeney et al., 1998), 10 items scored on a 4-point scale
Consequences of CB-PTSD : Relationship satisfaction (Mother) | 12 months postpartum
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Consequences of CB-PTSD : Relationship satisfaction (Partner) | 12 months postpartum
  Relationship assessment scale (RAS; Saramago et al., 2021), 7 items scored on a 5-point scale
Consequences of CB-PTSD : Coparenting (Mother) | 12 months postpartum
  Coparenting Relationship Scale (CRS; Favez et al., 2021), 35 items scored on a 7-point scale
Consequences of CB-PTSD : Coparenting (Partner) | 12 months postpartum
  Coparenting Relationship Scale (CRS; Favez et al., 2021), 35 items scored on a 7-point scale
Consequences of CB-PTSD : Support from neighborhood (Mother) | 12 months postpartum
  Perceived Neighborhood Social Cohesion (P-NSC; Dupuis et al., 2017), 9 items scored on a 7-point scale
Consequences of CB-PTSD : Support from neighborhood (Partner) | 12 months postpartum
  Perceived Neighborhood Social Cohesion (P-NSC; Dupuis et al., 2017), 9 items scored on a 7-point scale
Consequences of CB-PTSD : Healthcare renunciation (Mother) | 12 months postpartum
  Healthcare renunciation, 3 items
Consequences of CB-PTSD : Healthcare renunciation (Partner) | 12 months postpartum
  Healthcare renunciation, 3 items

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, Principal Investigator — UNIL-CHUV
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be available upon request

REFERENCES:
- [Derived] Chanvrier H, Rattaz V, Offredi V, Dupuis M, Horsch A. Swiss cohort on Traumatic Childbirth and Health (SwiTCH): protocol for a prospective, population-based cohort study on parents' mental health from pregnancy to one year postpartum. BMJ Open. 2024 Jan 30;14(1):e080557. doi: 10.1136/bmjopen-2023-080557. PMID 38296274